CLINICAL TRIAL: NCT03591172
Title: Assessment of Implementing Nano-technology in the Irrigation Protocol of One Step Revascularization For Necrotic Mature Teeth
Brief Title: Using Three Different Final Irrigants and Showing Their Effects on the Success of Revascularization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Ahmed Nassar, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEBD_CU_2018_05_29
Record Dates: First submitted 2018-06-26; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-05

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Propolis; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- propolis (Experimental): natural antibacterial, anti-inflammatory irrigation solution
  Interventions: Drug: Propolis
- Nano-propolis (Experimental): natural antibacterial, anti-inflammatory irrigation solution
  Interventions: Drug: Nano-propolis
- saline (Active Comparator): sodium chloride irrigation solution
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Propolis — Using propolis as a final irrigation in revascularization
  Other Names: natural irrigant
  Arms: propolis
Drug: Nano-propolis — Using Nano-propolis as a final irrigation in revasculariztion
  Other Names: Natural irrigant
  Arms: Nano-propolis
Drug: saline — Using saline as a final irrigation in revasculariztion
  Other Names: sodium chloride
  Arms: saline

SUMMARY:
this study will assess different irrigating materials on the success revascularization of necrotic mature teeth associated with PRF.

DETAILED DESCRIPTION:
Nano-propolis and Propolis will be used as final endodontic irrigants and will be compared to saline in Revascularization of necrotic mature teeth.

ELIGIBILITY:
Inclusion Criteria:

* mature teeth.
* teeth with periapical periodontitis.
* Maxillary anterior teeth
* Patients should be free from any systemic disease
* Patients who will agree to the consent and will commit to follow-up period.

Exclusion Criteria:

* Patients with immature roots.
* Patients with any systemic disease that may affect normal healing.
* Patients with swelling. .Pregnant females. .Patients who could/would not participate in a 1-year follow-up. .Patients with fistula. .Patients with old age. .Teeth with periodontal involvement. .Teeth with vertical root fractures. .Non-restorable teeth.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
post-operative pain: Visual analogue scale | 1 year
  post-operative pain evaluated using Visual analogue scale , 0 no pain, 10 severe pain.

SECONDARY OUTCOMES:
periapical healing | 1 year
  evaluated radiographically
sensitivity | 1 year
  electric pulp tester
survival | 1 year
  clinical evaluation